CLINICAL TRIAL: NCT05066711
Title: A Prospective, Multicenter Study Evaluating the Safety and Performance of the NuVasive® ACP System for the Treatment of Patients With Pathologic Conditions of the Cervical Spine
Brief Title: NuVasive® ACP System Study
Status: Enrolling by invitation | Type: Observational
Sponsor: NuVasive (Industry)
Responsible Party: Sponsor
Organization: Globus Medical Inc (Industry)
Other Study IDs: NUVA.ACP0721
Record Dates: First submitted 2021-09-23; First posted 2021-10-04 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Cervical Spondylosis; Cervical Radiculopathy; Cervical Myelopathy; Cervical Disc Disease; Cervical Stenosis; Cervical Disc Herniation; Cervical Spine Disease
Keywords: Spine surgery
MeSH Terms: conditions — Spondylosis; Radiculopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- ACP System

SUMMARY:
The primary objective of this study is to evaluate the safety and performance of anterior cervical spine surgery using the NuVasive anterior cervical plate (ACP) System as measured by reported complications, radiographic outcomes, and patient-reported outcomes (PROs).

DETAILED DESCRIPTION:
This study is a prospective, uncontrolled, multicenter study to evaluate the safety and performance of the NuVasive ACP System in patients who undergo anterior cervical spine surgery. Consecutive patients at a given site who meet eligibility requirements will be asked to consent to participate in the study. These patients will present with pathologic conditions in the cervical spine that are amenable to surgical treatment and will be screened prior to study enrollment. Once enrolled in the study, subjects will undergo anterior cervical spine surgery using the NuVasive ACP System based on the surgeon's standard of care. At least 75 subjects will be enrolled and will be followed for 24 months after the surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are ≥18 years of age at the time of consent
2. Have planned anterior cervical (C2 to C7) spine surgery using the NuVasive ACP System in conjunction with a NuVasive interbody implant or vertebral body replacement device (VBR), or a structural bone allograft spacer, for treatment of any of the following conditions:

   1. degenerative disc disease, as defined by neck pain of discogenic origin with degeneration of the disc confirmed by patient history and radiographic studies
   2. trauma (including fractures)
   3. tumors involving the cervical spine
   4. cervical spinal deformity (kyphosis, lordosis, or scoliosis)
   5. failed previous cervical fusion(s) (e.g., pseudoarthrosis)
   6. cervical spondylolisthesis
   7. cervical spinal stenosis
3. Able to undergo surgery based on physical exam, medical history, and surgeon judgment
4. Understands the conditions of enrollment and is willing to sign an informed consent form to participate in the study

Exclusion Criteria:

1. Procedures performed with interbody implants with integrated vertebral body screw(s)
2. Patient is involved in active litigation relating to the spine (worker's compensation claim is allowed if it is not contested)
3. Use of bone growth stimulators postoperatively
4. Active smoking within 6 weeks of surgery
5. Patient has known sensitivity to materials implanted
6. Systemic or local infection (latent or active) or signs of local inflammation
7. Patient has inadequate bone stock or quality, or a physical or medical condition that would prohibit beneficial surgical outcome based on surgeon judgment
8. Pregnant, or plans to become pregnant
9. Patient is a prisoner
10. Patient is participating in another clinical study that would confound study data

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The Enrolled Population will include all subjects who meet the criteria for enrollment, specifically, those subjects who:
  * Satisfied the inclusion and exclusion criteria,
  * Signed the informed consent, and
  * Underwent the surgical procedure, as defined in this protocol. Subjects not meeting any of these criteria will not be considered enrolled in the study, and therefore not included in any study population or analysis.
  The Evaluable Populations will include all subjects who:
  * Were included in the Enrolled Populations,
  * Completed the study, and
  * Had no major protocol deviations. If there are no major protocol deviations and all subjects complete the study, then an Evaluable Population will not be used.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2022-05-22 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Complications NuVasive ACP System | 24 months
  Rate of complications (i.e., safety) attributable to use of the NuVasive ACP System
Radiographic Success | 24 months
  Proportion of subjects with radiographic success at:
  1. Latest time point available for patients undergoing surgery to treat advanced stage tumors
  2. 24 months postoperative for subjects undergoing surgery to treat instabilities, traumatic spinal fractures, failed previous fusions, or degenerative disease

SECONDARY OUTCOMES:
Clinical Outcome Success | 24 months
  Percentage of subjects meeting minimal clinically important difference (MCID) and/or substantial clinical benefit (SCB) thresholds for each PRO: neck and arm pain (measured by visual analog scale (VAS)), disability (measured by neck disability index (NDI)), and overall physical and mental health (measured by PROMIS-10)
Rate of Postoperative Dysphagia | 24 months
  Rate of postoperative dysphagia as measured by the Eating Assessment Tool (EAT-10)
Rate of complications attributable to the use of NuVasive instruments, implants, or technologies | 24 months
  Rate of complications attributable to the use of NuVasive instruments, implants, or technologies

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Malone, MS, Study Director — Globus Medical Inc
Locations (3):
- United States (3):
  - Duly Health and Care, Naperville, Illinois
  - Columbia Orthopedic Group Research, Columbia, Missouri
  - Atlantic Brain and Spine, Wilmington, North Carolina